CLINICAL TRIAL: NCT01368978
Title: Evaluation of the Effect of lnsuPatch on the Pharmacokinetic and Pharmacodynamic Properties of Rapid-Acting Insulin Analogs Given as a Bolus by Continuous Subcutaneous Insulin Infusion (CSII)
Brief Title: Pediatric Diabetics Type 1 Using InsuPatch
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Insuline Medical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: G090175
Record Dates: First submitted 2010-12-21; First posted 2011-06-08 (Estimated); Last update posted 2014-09-05 (Estimated); Status verified 2012-05

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: TIDM
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test (with the InsuPatch device) (Experimental): Device use
  Interventions: Device: InsuPatch
- Control (without the InsuPatch device) (No Intervention)

INTERVENTIONS:
Device: InsuPatch — device which apply local heating at 38.5 degrees Celsius to the vicinity of the subcutaneous insulin infusion insertion site.
  Arms: Test (with the InsuPatch device)

SUMMARY:
This study is a prospective, single-center, open label, randomized; two-arms cross over study.

This is the test protocol for the InsuPatch device, whose purpose is to improve insulin delivery into the blood when the insulin is infused using an insulin-infusion pump by controlled heating of the area surrounding the point of infusion.

DETAILED DESCRIPTION:
Twenty(20) type 1 children with Type 1 Diabetics Mellitus (TIDM) who are meeting the inclusion/exclusion criteria as outlined below and who provide written Informed Consent will be enrolled in the study.

The study will consist of an outpatient enrollment visit and two admissions(One clamps with the InsuPatch and one clamp without the InsuPatch) . Each Subject will thus serve as his/her own control.

ELIGIBILITY:
Inclusion Criteria:

1. Age 12-17 (inclusive)
2. Clinical diagnosis of T1DM at least one year's duration
3. On CSII therapy for at least three months
4. Hemoglobin A1c(HBA1C) values below 10% and above 6.5%
5. Minimum weight requirements of at least 37.9 Kg.
6. Ability to comprehend written and spoken English
7. Body Mass Index z-score below 90%

Exclusion Criteria:

1. Celiac disease, gastroparesis, or other gastrointestinal disorder associated with alerted carbohydrate absorption or intestinal motility.
2. Medication besides insulin known to alter blood glucose, gastric motility, or intestinal carbohydrate absorption
3. Female subjects of reproductive potential who are pregnant or breast feeding
4. Inability to comprehend written and spoken English
5. Any other condition, which in the judgment of the investigators, would interfere with the subject's or parents' ability to provide informed consent or the investigator's ability to perform the study.
6. Hematocrit below 35 or serum potassium below 3.4 (confirmed by two samples)

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 27 (Actual)
Dates: Start 2009-12; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Efficacy | one year
  Insulin will be taken during the clamp and will be measured for concentration.The concentration of insulin during the first hour will be compared between the two arms for efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Eda Cengiz, MD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States